CLINICAL TRIAL: NCT00220324
Title: Prospective, Multicenter, Open-label, Uncontrolled Study to Investigate the Contraceptive Efficacy, Bleeding Patterns, and Safety of an Oral Contraceptive Containing 0.03 mg Ethinylestradiol and 0.125 mg Levonorgestrel (SH D00342A) Applied for 13 Cycles to Healthy Female Volunteers
Brief Title: Pearl Index Study With Low Dose Combined Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 91313; 307987 (Other: Other company ID)
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — Ethinyl Estradiol-Norgestrel Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Minisiston (SH D00342A)

INTERVENTIONS:
Drug: Minisiston (SH D00342A) — Daily oral administration in 21 days per cycle, followed by a 7-day pill-free interval

SUMMARY:
The purpose of this study is to investigate the contraceptive efficacy, bleeding pattern, and safety of SH D00342A. Subjects participating in the study will be treated with an oral contraceptive pill containing 0.03 mg ethinylestradiol and 0.125 mg levonorgestrel.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women requiring contraception

Exclusion Criteria:

* Pregnant or lactating women, history or suspicion of hormone dependent tumor or any other conditions which forbid the participation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 840 (Actual)
Dates: Start 2004-02; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Unadjusted Pearl Index | After 13 cycles of intake

SECONDARY OUTCOMES:
Adjusted Pearl Index | After 13 cycles of intake
Cumulative pregnancy rate | After 13 cycles of intake
Bleeding pattern | After 13 cycles of intake
Cycle control | After 13 cycles of intake

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Germany (13):
  - Hanover, Lower Saxony
  - Dresden, Saxony
  - Großpösna, Saxony
  - Leipzig, Saxony
  - Aschersleben, Saxony-Anhalt
  - Burg, Saxony-Anhalt
  - Egeln, Saxony-Anhalt
  - Halberstadt, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Suhl, Thuringia
  - Weida, Thuringia